CLINICAL TRIAL: NCT05637892
Title: A Multi-center Cohort Study of Hydatidiform Mole
Brief Title: A Cohort Study of Hydatidiform Mole
Status: Not yet recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20220312-R
Record Dates: First submitted 2022-11-01; First posted 2022-12-06 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Hydatidiform Mole
MeSH Terms: conditions — Hydatidiform Mole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect blood, and tissue samples from patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is a prospective observational study with no intervention

SUMMARY:
The purpose of this study is to construct a cohort for the hydatidiform mole.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients who meet the eligibility requirements will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with hydatidiform mole (including: complete hydatidiform mole/partial hydatidiform mole; one of twins with hydatidiform mole; ectopic pregnancy hydatidiform mole; macroscopic or microscopic hydatidiform changes indicating early complete or partial hydatidiform mole can not be excluded; atypical placental site nodule) for the first time;
2. Age 13-55 years old;
3. Obtain informed consent and sign an informed consent form

Exclusion Criteria:

1. Patients who are unable to cooperate with the investigation such as mental disorders or cognitive impairment
2. No histopathology diagnosis;
3. Patients with other malignancies

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Outpatient or inpatient patients in women's hospital school medicine of zhejiang university and other cooperative hospitals (including tongji hosptial, tongji medical college of hust, qilu hosptial of shandong university, Sun Yat-sen university cancer center) were inclued in this cohort study if the patients met the eligibility requirements and agreed to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Malignant trophoblastic tumor | 4.5 years
  Patients with hydatidiform mole develop malignant trophoblastic tumor. The Federation of International of Gynecologists and Obstetricians criteria for diagnosis of postmolar gestational trophoblastic neoplasia were as follows: (1) when the plateau of human chorionic gonadotrophin (hCG) lasts for four measurements over a period of 3 weeks or longer; that is, days 1, 7, 14, 21; (2) when there is a rise in hCG for three consecutive weekly measurements over at least a period of 2 weeks or more; days 1, 7, 14; (3) If there is a histologic diagnosis of choriocarcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Lv, PhD, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University

IPD SHARING:
Plan to Share IPD: No